CLINICAL TRIAL: NCT03559257
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Galcanezumab in Adults With Treatment-Resistant Migraine - the CONQUER Study
Brief Title: A Study of Galcanezumab (LY2951742) in Adults With Treatment-Resistant Migraine
Acronym: CONQUER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16670; I5Q-MC-CGAW (Other: Eli Lilly and Company); 2018-000600-42 (EudraCT Number)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2019-10

CONDITIONS: Migraine
Keywords: prevention; prophylaxis; headache; treatment-resistant; treatment resistant
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Galcanezumab (Experimental): Galcanezumab administered subcutaneously (SC).
  Interventions: Drug: Galcanezumab
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab — Administered SC.
  Other Names: LY2951742
  Arms: Galcanezumab
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of galcanezumab in people with treatment-resistant episodic or chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of migraine or chronic migraine.
* History of migraine headaches at least 1 year prior to screening, with onset prior to age 50.
* History of at least 4 migraine headache days and at, with at least 1 headache-free day per month on average within the past 3 months.
* Have documentation of 2 to 4 migraine preventive medication category failures due to inadequate efficacy or tolerability, in the past 10 years.

Exclusion Criteria:

* Are currently enrolled in or have participated within the last 30 days or within 5 half-lives (whichever is longer) in a clinical trial involving an investigational product.
* Current use or prior exposure to galcanezumab or another calcitonin gene-related peptide (CGRP) antibody.
* History of persistent daily headache, cluster headache or migraine subtypes including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, and migraine with brainstem aura (basilar-type migraine).
* Pregnant or nursing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (69):
- United States (18):
  - 21st Century Neurology, Phoenix, Arizona
  - Medical Center for Clinical Research, San Diego, California
  - Sensible Healthcare, Ocoee, Florida
  - University of South Florida, Tampa, Florida
  - Renstar Medical Research, Wesley Chapel, Florida
  - Boston Clinical Trials, Boston, Massachusetts
  - Michigan Head, Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Healthy Perspectives Innovative Mental Health Services, PL, Nashua, New Hampshire
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Rochester Clinical Research, Inc., Rochester, New York
  - PharmQuest, Greensboro, North Carolina
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - Foothill Family Clinic, Salt Lake City, Utah
  - Health Research of Hampton Roads Inc, Newport News, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Belgium (3):
  - Algemeen Ziekenhuis St Jan Brugge, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Canada (3):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - DIEX Recherche Sherbrooke, Inc, Sherbrooke, Quebec
- Czechia (6):
  - Clintrial, s.r.o., Prague, Hl. M. Praha
  - Neurologicka ambulance, Neurologie Brno s.r.o., Brno
  - Brain-Soultherapy s.r.o, Kladno
  - DADO MEDICAL, s.r.o., Prague
  - Neurologicka ordinace, Prague
  - Institut Neuropsychiatricke Pece, Prague
- France (3):
  - CHRU de Lille- Hôpital Roger Salengro, Lille, Cedex
  - Hôpital de Cimiez, Nice
  - CHU St Etienne Hopital Nord, Saint-Etienne
- Germany (5):
  - DRK-Kliniken Nordhessen, Kassel, Hesse
  - Praxis Dr. Philipp Stude, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Jena, Jena, Thuringia
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Essen, Essen
- Hungary (3):
  - Valeomed Kft., Esztergom, Komárom-Esztergom
  - SE Neurologiai Klinika, Budapest
  - Orszagos Idegtudomanyi Intezet, Budapest
- Japan (12):
  - Higashi Sapporo Neurology and Neurosurgery Clinic, Sapporo, Hokkaido
  - Medical corporation Shinmatsudakai Atago Hospital, Kochi, Kochi
  - Sendai Headache and Neurology Clinic, Sendai, Miyagi
  - Takase internal medicine clinic, Toyonaka-shi, Osaka
  - Dokkyo Medical University Hospital, Shimotsuga-Gun, Tochigi
  - Fukuuchi Pain Clinic, Shinjuku-ku, Tokyo
  - Shimoda Neurology Clinic, Tottori-shi, Tottori
  - Doi Clinic Internal Medicine Neurology, Hiroshima
  - Tanaka neurosurgical clinic, Kagoshima
  - Tatsuoka Neurology Clinic, Kyoto
  - Tominaga Hospital, Osaka
  - Ooba Clinic for Neurosurgery & Headache, Ōita
- Netherlands (2):
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Isala Klinieken, Zwolle
- Instituto de Neurologia Dra. Ivonne Fraga, San Juan, PR, Puerto Rico
- South Korea (4):
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hosp, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (6):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques De Valdecilla, Santander, Cantabria
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario La Fe de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- United Kingdom (3):
  - Hull Royal Infirmary, Hull, East Yorkshire
  - Kings College Hospital, London, Greater London
  - St Thomas's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Ford JH, Ye W, Ayer DW, Mi X, Bhandari S, Buse DC, Lipton RB. Validation and meaningful within-patient change in work productivity and activity impairment questionnaire (WPAI) for episodic or chronic migraine. J Patient Rep Outcomes. 2023 Apr 4;7(1):34. doi: 10.1186/s41687-023-00552-4. PMID 37016181
- [Derived] Ailani J, Andrews JS, Tockhorn-Heidenreich A, Wenzel R, Rettiganti M. Effect of Galcanezumab on Total Pain Burden in Patients Who Had Previously Not Benefited from Migraine Preventive Medication (CONQUER Trial): A Post Hoc Analysis. Adv Ther. 2022 Oct;39(10):4544-4555. doi: 10.1007/s12325-022-02233-y. Epub 2022 Aug 5. PMID 35930126
- [Derived] Ailani J, Kuruppu DK, Rettiganti M, Oakes T, Schroeder K, Wietecha L, Port M, Blumenfeld AM. Does "wearing off" of efficacy occur in galcanezumab-treated patients at the end of the monthly treatment cycle? Post hoc analyses of four phase III randomized trials. Headache. 2022 Feb;62(2):198-207. doi: 10.1111/head.14257. Epub 2022 Jan 25. PMID 35076090
- [Derived] Tepper SJ, Ailani J, Ford JH, Nichols RM, Li LQ, Kemmer P, Hand AL, Tockhorn-Heidenreich A. Effects of Galcanezumab on Health-Related Quality of Life and Disability in Patients with Previous Failure of 2-4 Migraine Preventive Medication Categories: Results from a Phase IIIb Randomized, Placebo-Controlled, Multicenter Clinical Trial (CONQUER). Clin Drug Investig. 2022 Mar;42(3):263-275. doi: 10.1007/s40261-021-01115-5. Epub 2022 Jan 18. PMID 35041159
- [Derived] Okonkwo R, Tockhorn-Heidenreich A, Stroud C, Paget MA, Matharu MS, Tassorelli C. Efficacy of galcanezumab in patients with migraine and history of failure to 3-4 preventive medication categories: subgroup analysis from CONQUER study. J Headache Pain. 2021 Sep 30;22(1):113. doi: 10.1186/s10194-021-01322-7. PMID 34592919
- [Derived] Reuter U, Lucas C, Dolezil D, Hand AL, Port MD, Nichols RM, Stroud C, Tockhorn-Heidenreich A, Detke HC. Galcanezumab in Patients with Multiple Previous Migraine Preventive Medication Category Failures: Results from the Open-Label Period of the CONQUER Trial. Adv Ther. 2021 Nov;38(11):5465-5483. doi: 10.1007/s12325-021-01911-7. Epub 2021 Sep 20. PMID 34542830
- [Derived] Citrome L, Sanchez Del Rio M, Dong Y, Nichols RM, Tockhorn-Heidenreich A, Foster SA, Stauffer VL. Benefit-Risk Assessment of Galcanezumab Versus Placebo for the Treatment of Episodic and Chronic Migraine Using the Metrics of Number Needed to Treat and Number Needed to Harm. Adv Ther. 2021 Aug;38(8):4442-4460. doi: 10.1007/s12325-021-01848-x. Epub 2021 Jul 15. PMID 34264500
- [Derived] Kuruppu DK, Tobin J, Dong Y, Aurora SK, Yunes-Medina L, Green AL. Efficacy of galcanezumab in patients with migraine who did not benefit from commonly prescribed preventive treatments. BMC Neurol. 2021 Apr 23;21(1):175. doi: 10.1186/s12883-021-02196-7. PMID 33892641
- [Derived] Schwedt TJ, Kuruppu DK, Dong Y, Standley K, Yunes-Medina L, Pearlman E. Early onset of effect following galcanezumab treatment in patients with previous preventive medication failures. J Headache Pain. 2021 Mar 25;22(1):15. doi: 10.1186/s10194-021-01230-w. PMID 33765912
- [Derived] Mulleners WM, Kim BK, Lainez MJA, Lanteri-Minet M, Pozo-Rosich P, Wang S, Tockhorn-Heidenreich A, Aurora SK, Nichols RM, Yunes-Medina L, Detke HC. Safety and efficacy of galcanezumab in patients for whom previous migraine preventive medication from two to four categories had failed (CONQUER): a multicentre, randomised, double-blind, placebo-controlled, phase 3b trial. Lancet Neurol. 2020 Oct;19(10):814-825. doi: 10.1016/S1474-4422(20)30279-9. Epub 2020 Sep 16. PMID 32949542
- See also: A Study of Galcanezumab (LY2951742) in Adults With Treatment-Resistant Migraine — https://www.lillytrialguide.com/en-US/studies/migraine/CGAW

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Galcanezumab 120mg: Participants received matching placebo every month for three months by subcutaneous injection (SC) during double blind treatment phase. Participants received initial loading dose of 240mg galcanezumab followed by 120mg every month for two months by SC injection during open label treatment period.
- Galcanezumab 120mg: Participants received initial loading dose of 240mg of galcanezumab followed by 120mg galcanezumab every month for two months by SC injection during double blind treatment period. Participants received 120mg of galcanezumab every month for three months by SC injection during open label treatment period.
Period: Double Blind Treatment Period
Arm/Group | Placebo/Galcanezumab 120mg | Galcanezumab 120mg
Started | 230 | 233
Received at Least One Dose of Study Drug | 230 | 232
Completed | 226 | 225
Not Completed | 4 | 8
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 1 | 4
Not completed — Lack of Efficacy | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Screen Failure | 0 | 1
Period: Open-label Treatment Period
Arm/Group | Placebo/Galcanezumab 120mg | Galcanezumab 120mg
Started | 225 (One participant who completed double blind period has withdrawn from the study.) | 224 (One participant who completed double blind period had discontinued due to adverse event.)
Completed | 215 | 217
Not Completed | 10 | 7
Not completed — Adverse Event | 1 | 4
Not completed — Lack of Efficacy | 3 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Galcanezumab 120mg | Galcanezumab 120mg | Total
Number analyzed (Participants) | 230 | 232 | 462
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.67 (12.33) | 45.87 (11.34) | 45.77 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 195 | 397
  Male | 28 | 37 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 31
  Not Hispanic or Latino | 174 | 172 | 346
  Unknown or Not Reported | 40 | 45 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 35 | 37 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 182 | 183 | 365
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 7 | 8 | 15
Monthly Migraine Headache Days [Mean (Standard Deviation); unit: Days] | 13.01 (5.73) | 13.44 (6.08) | 13.23 (5.91)

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days
Description: Migraine Headache Day (MHD): A calendar day on which a migraine headache or probable migraine headache occurred.
  Overall mean is derived from the average of months 1 to 3 from mixed model repeated measures (MMRM) model. Least square (LS) Mean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 3
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline value.
Measure: Least Squares Mean (Standard Error); unit: Days
Groups:
- Placebo - Double-Blind Treatment Phase: Participants received matching placebo every month for three months by SC injection.
- Galcanezumab 120mg - Double-Blind Treatment Phase: Participants received initial loading dose of 240 milligrams (mg) of galcanezumab followed by 120mg Galcanezumab every month for two months by SC injection.
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 228 | 230
Days | -1.02 (0.32) | -4.14 (0.32)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSMean Difference = -3.12, 95% CI 2-sided [-3.92 to -2.32], Standard Error of Mean 0.41

2. Secondary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days in Participants With Episodic Migraine
Description: MHD: A calendar day on which a migraine headache or probable migraine headache occurred.
  Overall mean is derived from the average of months 1 to 3 from MMRM model. Least square (LS) Mean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 3
Population: All randomized episodic migraine participants who received at least one dose of study drug and had baseline and at least one post baseline value.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 132 | 137
Days | -0.31 (0.34) | -2.88 (0.34)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSMean Difference = -2.57, 95% CI 2-sided [-3.41 to -1.72], Standard Error of Mean 0.43

3. Secondary Outcome: Percentage of Participants With ≥50% Reduction From Baseline in Monthly Migraine Headache Days
Description: MHD: A calendar day on which a migraine headache or probable migraine headache occurred.
  Overall mean percentage across months 1 through 3 of patients with at least a 50% reduction in monthly MHDs from baseline using a categorical pseudo likelihood-based repeated measures model for binary responder indicator with fixed, categorical effects of treatment, month, treatment by month, and continuous, fixed covariate of baseline monthly MHD.
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 228 | 230
Percentage of Participants | 13.3 [10.2 to 17.3] | 37.7 [32.9 to 42.8]
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, pseudo likelihood-based repeated measure; Odds Ratio (OR) = 3.935, 95% CI 2-sided [2.719 to 5.693]

4. Secondary Outcome: Percentage of Participants With Episodic Migraine With ≥50% Reduction From Baseline in Monthly Migraine Headache Days
Description: as for outcome 3
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 132 | 137
Percentage of Participants | 17.1 [12.7 to 22.7] | 41.8 [35.7 to 48.1]
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, Pseudo likelihood-based repeated measure; Odds Ratio (OR) = 3.481, 95% CI 2-sided [2.252 to 5.381]

5. Secondary Outcome: Mean Change From Baseline in the Role Function-Restrictive Domain Score of the Migraine-Specific Quality of Life Questionnaire Version 2.1 (MSQ v2.1)
Description: MSQ v2.1 is a health status instrument, with a 4-week recall period, developed to address physical and emotional limitations of specific concern to individuals with migraine. Addressing the impact of migraine on work or daily activities, relationships with family & friends, leisure time, productivity, concentration, energy, tiredness & feelings. It consists of 14 items that address 3 domains:(1) Role Function-Restrictive (items 1-7);(2) Role Function- Preventive (items 8-11);&(3) Emotional Function (items 12-14).Response options range from "none of the time" (value 1) to "all of the time" (value 6),& are reverse-recoded (value 6 to 1) before the domain scores are calculated. Total raw scores for each domain is the sum of the final item value for all of the items in that domain. After the total raw score is computed for each domain, they are transformed to a 0-100 scale with higher scores indicating a better health status & a positive change in scores reflecting functional improvement.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had a post baseline value at Month 3.
  LS Mean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, and baseline by month as fixed effects.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 222 | 223
score on a scale | 10.68 (1.34) | 23.21 (1.35)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSMean Difference = 12.53, 95% CI 2-sided [9.19 to 15.87], Standard Error of Mean 1.70

6. Secondary Outcome: Mean Change From Baseline in the Role Function-Restrictive Domain Score of the Migraine-Specific Quality of Life Questionnaire Version 2.1 (MSQ v2.1) in Participants With Episodic Migraine
Description: as for outcome 5
Time Frame: Baseline, Month 3
Population: All randomized episodic migraine participants who received at least one dose of study drug and had a post baseline value at Month 3. LS Mean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, and baseline by month as fixed effects.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 127 | 135
score on a scale | 11.88 (1.80) | 23.39 (1.79)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSMean Difference = 11.51, 95% CI 2-sided [7.14 to 15.89], Standard Error of Mean 2.22

7. Secondary Outcome: Percentage of Participants With Episodic Migraine With ≥75% Reduction From Baseline in Monthly Migraine Headache Days
Description: MHD: A calendar day on which a migraine headache or probable migraine headache occurred.
  Overall mean percentage across months 1 through 3 of patients with at least a 75% reduction in monthly MHDs from baseline using a categorical pseudo likelihood-based repeated measures model for binary responder indicator with fixed, categorical effects of treatment, month, treatment by month, and continuous, fixed covariate of baseline monthly MHD.
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 132 | 137
Percentage of Participants | 3.7 [1.6 to 8.2] | 18.4 [13.9 to 23.9]
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p = 0.0001, Pseudo likelihood-based repeated measure; Odds Ratio (OR) = 5.878, 95% CI 2-sided [2.374 to 14.554]

8. Secondary Outcome: Percentage of Participants With Episodic Migraine With 100% Reduction From Baseline in Monthly Migraine Headache Days
Description: MHD: A calendar day on which a migraine headache or probable migraine headache occurred.
  Overall mean percentage across months 1 through 3 of patients with 100% reduction in monthly MHDs from baseline using a categorical pseudo likelihood-based repeated measures model for binary responder indicator with fixed, categorical effects of treatment, month, treatment by month, and continuous, fixed covariate of baseline monthly MHD.
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 132 | 137
Percentage of Participants | 0.00 [0.00 to 0.00] | 7.7 [4.7 to 12.3]
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, Pseudo likelihood-based repeated measure; Odds Ratio (OR) = 999.999, 95% CI 2-sided [548.706 to 999.999] — Estimated value and upper bound are >999.999

9. Secondary Outcome: Percentage of Participants With ≥75% Reduction From Baseline in Monthly Migraine Headache Days
Description: as for outcome 7
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 228 | 230
Percentage of Participants | 3.3 [1.7 to 6.3] | 14.5 [10.9 to 19.0]
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, pseudo likelihood-based repeated measure; Odds Ratio (OR) = 5.012, 95% CI 2-sided [2.352 to 10.679]

10. Secondary Outcome: Percentage of Participants With 100% Reduction From Baseline in Monthly Migraine Headache Days
Description: as for outcome 8
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 228 | 230
Percentage of Participants | 0.000 [0.000 to 0.000] | 4.9 [2.8 to 8.6]
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, Pseudo likelihood-based repeated measure; Odds Ratio (OR) = 999.99, 95% CI 2-sided [999.99 to 999.99] — Point estimate, upper limit and lower limit are >999.99

11. Secondary Outcome: Overall Mean Change From Baseline in the Number of Monthly Days With Acute Headache Medication Use
Description: Overall mean is derived from the average of months 1 to 3 from Mixed model repeated measures (MMRM) model. Least square (LS) Mean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 228 | 230
Days | -0.80 (0.31) | -4.19 (0.32)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSMean Difference = -3.40, 95% CI 2-sided [-4.14 to -2.65], Standard Error of Mean 0.38

12. Secondary Outcome: Overall Mean Change From Baseline in the Number of Monthly Headache Days
Description: Headache Day: A calendar day on which any type of headache occurred (including migraine, probable migraine, and non-migraine headache).
  Overall mean is derived from the average of months 1 to 3 from MMRM model. Least square (LS) Mean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 228 | 230
Days | -1.05 (0.36) | -4.18 (0.35)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSMean Difference = -3.13, 95% CI 2-sided [-3.96 to -2.29], Standard Error of Mean 0.42

13. Secondary Outcome: Mean Change From Baseline in the Migraine Disability Assessment Test (MIDAS) Total Score
Description: The MIDAS is a participant-rated scale which was designed to quantify headache-related disability over a 3-month period. This instrument consists of five items that reflect the number of days reported as missed or with reduced productivity at work or home, and the number of days of missed social events. Each item has a numeric response range from 0 to 90 days, if days are missed from work or home they are not counted as days with reduced productivity at work or home. The numeric responses are summed to produce a total score ranging from 0 to 270, in which a higher value is indicative of more disability. LS mean was calculated using analysis of covariance (ANCOVA) with last observation carried forward (LOCF), with baseline, pooled country, baseline migraine frequency category, and treatment as fixed effects.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had a post baseline value at Month 3.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 225 | 228
score on a scale | -3.295 (3.2834) | -21.097 (3.3164)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, ANCOVA

14. Secondary Outcome: Mean Change From Baseline in the 4-item Migraine Interictal Burden Scale (MIBS-4)
Description: MIBS-4 is a self-administered scale that measures the burden related to headache in the time between attacks. The instrument consists of 4 items that address disruption at work and school, diminished family and social life, difficulty planning, and emotional difficulty. The questionnaire specifically asks about the effect of the disease over the past 4 weeks on days without a headache attack. Response options include: don't know/not applicable (0), never (0), rarely (1), some of the time (2), much of the time (3), or most or all of the time (3). Each responses associated numerical score are summed across all 4 items resulting in a total score ranging from 0 to 12, and the level of interictal burden being categorized into the following: 0 for none, 1-2 mild, 3-4 moderate, and >5 severe. LS mean was calculated using MMRM model with fixed effects of treatment, pooled country, baseline migraine frequency category, month, treatment by month as fixed effects.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had a post baseline value at Month 3.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 222 | 223
score on a scale | -0.78 (0.21) | -1.83 (0.21)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LSMean Difference = -1.06, 95% CI 2-sided [-1.58 to -0.54], Standard Error of Mean 0.27

15. Secondary Outcome: Mean Change From Baseline in the Work Productivity and Activity Impairment Questionnaire (WPAI)
Description: The WPAI Questionnaire is a patient-reported instrument developed to measure the impact on work productivity and regular activities attributable to a specific health problem (migraine). Recall period is the past 7 days. It contains 6 items that measure: 1) employment status, 2) hours missed from work due to the specific health problem, 3) hours missed from work for other reasons, 4) hours actually worked, 5) degree health affected productivity while working, and 6) degree health affected productivity in regular unpaid activities. Four scores are calculated from the responses to these 6 items: absenteeism, presenteeism, work productivity loss, and activity impairment. Scores are calculated as impairment percentages (0-100%), with higher numbers indicating greater impairment and less productivity, i.e, worse outcomes. LS mean was calculated using ANCOVA with LOCF with baseline, pooled country, baseline migraine frequency category, and treatment as fixed effects.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had a post baseline value at Month 3.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 225 | 227
score on a scale
  Activity Impairment | -8.644 (1.9195) | -20.713 (1.9537)
  Absenteeism: number analyzed (Participants) | 145 | 148
  Absenteeism | -2.900 (1.2436) | -4.224 (1.2929)
  Presenteeism: number analyzed (Participants) | 141 | 147
  Presenteeism | -2.564 (2.3222) | -12.504 (2.3705)
  Work Impairment: number analyzed (Participants) | 145 | 148
  Work Impairment | -3.457 (2.4098) | -14.307 (2.5148)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Activity Impairment; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Absenteeism; Test type: Superiority; p = 0.3880, ANCOVA
Statistical Analysis 3: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Presenteeism; Test type: Superiority; p = 0.0004, ANCOVA
Statistical Analysis 4: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Work impairment; Test type: Superiority; p = 0.0003, ANCOVA

16. Secondary Outcome: Mean Change From Baseline in the Patient Global Impression of Severity (PGI-S)
Description: The PGI-S is a patient-rated instrument that measures illness severity. For this study, the patient was instructed as follows: "Considering migraine as a chronic condition, how would you rate your level of illness?" The PGI-S includes a range of possible responses, from 1 ("normal, not at all ill") to 7 ("extremely ill"). LS mean was calculated using ANCOVA with LOCF with baseline, pooled country, baseline migraine frequency category, and treatment as fixed effects.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had a post baseline value at Month 3.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 225 | 228
score on a scale | -0.283 (0.0863) | -0.664 (0.0873)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p = 0.0003, ANCOVA

17. Secondary Outcome: Mean Change From Baseline in the European Quality of Life Questionnaire 5 Dimensions 5 Levels (EQ-5D-5L) - Health State Index (US)
Description: EQ-5D-5L is a 2-part questionnaire that assesses general health status for 'today'. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using country-specific algorithms, with scores ranging from less than 0 (where zero is a health state equivalent to death; negative values are valued as worse than dead) to 1 (perfect health). Index values were calculated using the US algorithm (-0.109 to 1). A higher score indicates better health state. LS mean was calculated using ANCOVA with LOCF with baseline, pooled country, baseline migraine frequency category, and treatment as fixed effects.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had a post baseline value at Month 3.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 225 | 227
score on a scale | -0.002 (0.0079) | 0.013 (0.0080)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p = 0.1267, ANCOVA

18. Secondary Outcome: Mean Change From Baseline in the European Quality of Life Questionnaire 5 Dimensions 5 Levels (EQ-5D-5L) - Health State Index (UK)
Description: EQ-5D-5L is a 2-part questionnaire that assesses general health status for 'today'. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using country-specific algorithms, with scores ranging from less than 0 (where zero is a health state equivalent to death; negative values are valued as worse than dead) to 1 (perfect health). Index values were calculated using the UK algorithm (-0.594 to 1). LS mean was calculated using ANCOVA with LOCF with baseline, pooled country, baseline migraine frequency category, and treatment as fixed effects.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had a post baseline value at Month 3.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 225 | 227
score on a scale | -0.001 (0.0109) | 0.017 (0.0110)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p = 0.1630, ANCOVA

19. Secondary Outcome: Mean Change From Baseline in the European Quality of Life Questionnaire 5 Dimensions 5 Levels (EQ-5D-5L) - VAS Score
Description: EQ-5D-5L is a 2-part questionnaire that assesses general health status 'today'. . The second part is assessed using a visual analog scale (VAS) on which the patient rates their perceived health state, ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine). LS mean was calculated using ANCOVA with LOCF with baseline, pooled country, baseline migraine frequency category, and treatment as fixed effects.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had a post baseline value at Month 3.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase
Number analyzed (Participants) | 225 | 227
mm | -0.086 (1.2916) | 3.376 (1.3080)
Statistical Analysis 1: Comparison: Placebo - Double-Blind Treatment Phase vs Galcanezumab 120mg - Double-Blind Treatment Phase; Test type: Superiority; p = 0.0277, ANCOVA

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Placebo/Galcanezumab 120mg - Open-Label Treatment Phase: Participants received initial loading dose of 240mg Galcanezumab followed by 120mg every month for two months by SC injection.
- Galcanezumab 120mg/Galcanezumab 120mg - Open-Label Treatment: Participants received 120mg of Galcanezumab every month for three months by SC injection.
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase | Placebo/Galcanezumab 120mg - Open-Label Treatment Phase | Galcanezumab 120mg/Galcanezumab 120mg - Open-Label Treatment
All-Cause Mortality (participants affected / at risk) | 0/230 | 0/232 | 0/225 | 0/224
Serious Adverse Events (participants affected / at risk) | 2/230 | 2/232 | 6/225 | 3/224
Other Adverse Events (participants affected / at risk) | 31/230 | 21/232 | 19/225 | 13/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Double-Blind Treatment Phase (N=230) | Galcanezumab 120mg - Double-Blind Treatment Phase (N=232) | Placebo/Galcanezumab 120mg - Open-Label Treatment Phase (N=225) | Galcanezumab 120mg/Galcanezumab 120mg - Open-Label Treatment (N=224)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0/202 (0) | 0/195 (0) | 0/197 (0) | 1/187 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Behcet's syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Double-Blind Treatment Phase (N=230) | Galcanezumab 120mg - Double-Blind Treatment Phase (N=232) | Placebo/Galcanezumab 120mg - Open-Label Treatment Phase (N=225) | Galcanezumab 120mg/Galcanezumab 120mg - Open-Label Treatment (N=224)
Injection site pain (General disorders) | 13 (30) | 5 (7) | 11 (19) | 5 (7)
Nasopharyngitis (Infections and infestations) | 21 (24) | 16 (17) | 11 (11) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03559257/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03559257/SAP_001.pdf